CLINICAL TRIAL: NCT00864656
Title: Comparative Study of Eyelid Position Interdependence in Involutional Ptosis Patients Submitted to 1, 2 or 4 Drops of 10% Phenylephrine
Brief Title: Eyelid Position Interdependence in Involutional Ptosis Patients Submitted to 10% Phenylephrine
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Suzana Matayoshi, Clinica Oftalmologica HCFMUSP
Other Study IDs: phenylephrine test
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Blepharoptosis
Keywords: adrenergic alpha-agonists; phenylephrine; drug effects; diagnostic use
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Patients submitted to application of 1 drop of 10% phenylephrine
- 2: Patients submitted to application of 2 drops of 10% phenylephrine
- 3: Patients submitted to application of 4 drops of 10% phenylephrine

SUMMARY:
The primary aim of this study is to quantify eyelid position changes in tested and opposite eyes in ptosis patients submitted to 1, 2 or 4 drops of 10% phenylephrine in one eye. The secondary objective is to correlate the eye dominance, severity and laterality of ptosis with eyelid position changes in these 3 groups.

DETAILED DESCRIPTION:
This is a prospective observational study conducted in involutional ptosis patients, which will be submitted to instillation of a single drop of 10% phenylephrine in one eye(Group 1), 2 drops (G2) or 4 drops ( G3).

Video camera will record the images of both eyes before and after drug application at 3, 10, 15 and 30 minutes. The images will be edited to analyze upper and lower lid height.

ELIGIBILITY:
Inclusion Criteria:

* Involutional blepharoptosis
* Upper Margin-reflex distance less or equal 2.0mm
* Good fixation and collaboration

Exclusion Criteria:

* Previous eyelid surgeries
* Use of adrenergic or sympathicomimetics drugs
* Myopathies
* Thyroid orbitopathy
* Non-controlled cardiovascular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Involutional blepharoptosis patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Upper lid height before and after phenylephrine test lower lid height before and after phenylephrine test | 3, 10, 15 and 30 minutes

SECONDARY OUTCOMES:
Scobee test to detect eye dominance | 15 minutes before 10% phenylephrine instillation

CONTACTS AND LOCATIONS:
Overall Officials: Suzana Matayoshi, MD, Principal Investigator — Opthalmology Dept.Sao Paulo University General Hospital
Locations (1):
- Ophthalmology Dept. University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Nunes TP, Matayoshi S. [Phenylephrine 10% eye drop action in the eyelid position in healthy subjects]. Arq Bras Oftalmol. 2008 Sep-Oct;71(5):639-43. doi: 10.1590/s0004-27492008000500006. Portuguese. PMID 19039456